CLINICAL TRIAL: NCT00670384
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose-Ranging Study of Sublingual Immunotherapy in Adults Sensitized to the Standardized Allergenic Extract, Short Ragweed (Ambrosia Artemisiifolia)
Brief Title: Phase 2 Study in Adults Sensitized to Short Ragweed
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding.
Sponsor: Antigen Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALI001-08
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Allergic Rhinitis
Keywords: SLIT; Immunotherapy; Short ragweed; SAR; Seasonal allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose Group A (Active Comparator): Standardized Allergenic Extract, Short Ragweed (Ambrosia artemisiifolia)
  Interventions: Biological: Standardized Allergenic Extract, Short Ragweed (Ambrosia artemisiifolia)
- Dose Group B (Active Comparator): Standardized Allergenic Extract, Short Ragweed (Ambrosia artemisiifolia)
  Interventions: Biological: Standardized Allergenic Extract, Short Ragweed (Ambrosia artemisiifolia)
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Standardized Allergenic Extract, Short Ragweed (Ambrosia artemisiifolia) — Sublingual drops
  Arms: Dose Group A; Dose Group B
Biological: Placebo — Sublingual drops
  Arms: Placebo

SUMMARY:
The purpose of this study is to identify an effective dose of allergen-specific immunotherapy for short ragweed (Ambrosia artemisiifolia) administered by an oral/sublingual route.

ELIGIBILITY:
Inclusion Criteria

* Male and female patients between the ages of 18 and 55 years (inclusive.
* Written informed consent to participate in the study.
* Documented allergy to short ragweed pollen as demonstrated by a positive epicutaneous skin test (wheal >3 mm) and symptoms of allergic rhinitis during the two previous short ragweed seasons.
* Female subjects of childbearing potential, defined as not surgically sterile or at least 2 years postmenopausal, must agree to use one of the following forms of contraception from screening through the 4 week follow-up period following the last dose of Clinical Trial Material (CTM): hormonal (oral, implant, or injection) begun >30 days prior to screening, barrier (condom, diaphragm with spermicide), Intrauterine Device (IUD), or vasectomized partner (6 months minimum).
* No clinically significant abnormal findings on the physical examination, with the exception of head, eyes, ears, nose and throat (HEENT) findings consistent with allergic rhinitis, medical history, or clinical laboratory results during screening which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results

Exclusion Criteria:

* Previous allergen immunotherapy (subcutaneous immunotherapy (SCIT), oral immunotherapy, sublingual immunotherapy (SLIT), or recombinant peptide) for short ragweed within 24 months of the Screening Visit.
* History of severe allergic reaction requiring medical intervention.
* Intolerance of or severe allergic reaction to previous immunotherapy (SCIT, oral immunotherapy, SLIT, or recombinant peptide).
* Allergy to any of the non-antigen ingredients in the study drug formulation, including, but not limited to, Food, Drug and Cosmetic (FD&C) Yellow #5, sodium chloride, sodium bicarbonate, and glycerine.
* History of asthma requiring daily medication.
* Subjects receiving anti-IgE monoclonal antibodies.
* Congenital immune deficiency or acquired immune suppression. Causes of acquired immune suppression may include, but are not limited to, systemic illnesses such as malignancy and infection, the use of medications such as corticosteroids and chemotherapeutic agents, and radiation therapy.
* History of organ transplant, hematologic malignancy, autoimmune disease, myocardial infarction, or congestive heart failure.
* History of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, psychiatric, or cardiovascular disease, or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Inability or unwillingness to stop using drugs that may inhibit the wheal-and-flare reaction or rhinitic response prior to the study and for the duration of dosing CTM (with the exception of protocol-specified rescue medications provided by the study site for use after Study Day 0).
* Inability or unwillingness to stop using drugs that may inhibit the ability to treat a severe allergic adverse event. This includes, but is not limited to: beta blockers such as atenolol (Tenormin), metoprolol (Lopressor, Toprol-XL) and propranolol (Inderal, Inderal LA) for 14 days prior to Study Day 0 and for the duration of the study
* Female subjects who are trying to conceive, are pregnant, or are lactating.
* Positive serum pregnancy test at screening or a positive human chorionic gonadotropin (HCG) urine test on Study Day 0 prior to administration of study drug for women of childbearing potential.
* Positive blood screen for HIV, Hepatitis B surface antigen (HbSAg), or Hepatitis C.
* History of alcohol or drug abuse within the year prior to the Screening Visit, or current evidence of substance dependence or abuse.
* Participation in a clinical trial or receipt of a non-FDA approved therapy within 30 days prior to the Screening Visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Average of Total Symptom Scores | 20 weeks